CLINICAL TRIAL: NCT05431530
Title: Assessment of Quality of Life After Low Anterior Resection or Visceral Peritoneal Stripping During cytOreDuctive surgerY for Advanced Ovarian Cancer Requiring Tumor Resection on the Rectosigmoid Colon: a Prospective Cohort Study
Brief Title: Assessment of Quality of Life After Low Anterior Resection During Cytoreductive Surgery for Advanced Ovarian Cancer
Acronym: LAPSODY
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LARS-1.0
Record Dates: First submitted 2022-06-19; First posted 2022-06-24 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Ovarian Cancer; Low Anterior Resection Syndrome; Quality of Life
MeSH Terms: conditions — Ovarian Neoplasms; Low Anterior Resection Syndrome | interventions — Cytoreduction Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ovarian cancer: Tumor involving rectosigmoid colon
  Interventions: Procedure: Cytoreductive surgery

INTERVENTIONS:
Procedure: Cytoreductive surgery — Cytoreductive surgery including resection of tumors involving rectosigmoid colon.

SUMMARY:
This study aims to evaluate the incidence of low anterior resection syndrome and quality of life after cytoreductive surgery for advanced ovarian cancer patients.

DETAILED DESCRIPTION:
In advanced ovarian cancer, 24-64% of patients require removal of tumors located in the rectum and sigmoid colon. In order to remove the tumor located in the rectum and sigmoid colon, low anterior resection (LAR) is performed to excise the rectum and sigmoid colon. All patients who underwent low anterior resection are at risk of developing low anterior resection syndrome, which presents symptoms such as frequent bowel movements, frequent defecation, and impaired stool control. Therefore, this study aims to evaluate the incidence of low anterior resection syndrome and quality of life after cytoreductive surgery for advanced ovarian cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Those with newly diagnosed ovarian cancer, fallopian tube cancer and primary peritoneal carcinomatosis who plan to undergo cytoreductive surgery and secondary cytoreductive surgery after neoadjuvant chemotherapy.
* Patients with PCDS or rectal and sigmoid coloni tumor invasion suspected on the preoperative image and need resection of the tumor and clinical FIGO stage IIIB or higher
* ECOG performance status : 0-2
* Age over 18

Exclusion Criteria:

* Patient who underwent low anterior resection in the past
* Past history of gastrointestinal malignant tumor except to ovarian cancer
* Patient who have colostomy
* Patient who underwent radiation therapy to abdominal or pelvic cavity
* ECOG performance status over 3
* Patient taking opioid analgesics
* Patient who have intellectual disability or dementia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: According to the existing literature report, 37.9% to 43.3% of cases of low anterior resection are expected to occur.
  Therefore, assuming that the major LARS incidence rate is 40%, and the number of subjects to estimate the incidence rate estimation precision (half of the 95% confidence interval width) within 10% is 93 patients. Considering the loss or death rate of 13.2% during follow-up within 1 year in our hospital, the number of subjects required is 108.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of major LARS after surgery | 12 months after LAR implementation
  Frequency of major LARS (corresponding to 30-42 points as a result of LARS questionnaire) 12 months after LAR implementation

SECONDARY OUTCOMES:
Incidence of major, minor LARS after visceral peritoneal stripping | 2weeks after surgery
  Incidence of major, minor LARS after visceral peritoneal stripping, not LAR
LARS severity | 2weeks before surgery, 2weeks after surgery(before adjuvant chemotherapy), 3,6,12,24 months after surgery
  LARS severity of before and after surgery(before adjuvant chemotherapy)
The fecal incontinency quality of life scale(FIQL) | 2weeks before surgery, 2weeks after surgery(before adjuvant chemotherapy), 3,6,12,24 months after surgery
  FIQL of before and after surgery
Bristol stool form scale | 2weeks before surgery, 2weeks after surgery(before adjuvant chemotherapy), 3,6,12,24 months after surgery
  Bristol stool form scale of before and after surgery
EORTC QLQ-Ov28 | 2weeks before surgery, 6,12,24 months after surgery
  EORTC QLQ-Ov28 of before and after surgery
EOTC QLQ-C30 | 2weeks before surgery, 6,12,24 months after surgery
  EOTC QLQ-C30 of before and after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hee Seung Kim, MD/PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aletti GD, Dowdy SC, Gostout BS, Jones MB, Stanhope CR, Wilson TO, Podratz KC, Cliby WA. Aggressive surgical effort and improved survival in advanced-stage ovarian cancer. Obstet Gynecol. 2006 Jan;107(1):77-85. doi: 10.1097/01.AOG.0000192407.04428.bb. PMID 16394043
- [Background] Bristow RE, Tomacruz RS, Armstrong DK, Trimble EL, Montz FJ. Survival effect of maximal cytoreductive surgery for advanced ovarian carcinoma during the platinum era: a meta-analysis. J Clin Oncol. 2002 Mar 1;20(5):1248-59. doi: 10.1200/JCO.2002.20.5.1248. PMID 11870167
- [Background] Chang SJ, Bristow RE. Evolution of surgical treatment paradigms for advanced-stage ovarian cancer: redefining 'optimal' residual disease. Gynecol Oncol. 2012 May;125(2):483-92. doi: 10.1016/j.ygyno.2012.02.024. Epub 2012 Feb 23. PMID 22366151
- [Background] Chen TY, Wiltink LM, Nout RA, Meershoek-Klein Kranenbarg E, Laurberg S, Marijnen CA, van de Velde CJ. Bowel function 14 years after preoperative short-course radiotherapy and total mesorectal excision for rectal cancer: report of a multicenter randomized trial. Clin Colorectal Cancer. 2015 Jun;14(2):106-14. doi: 10.1016/j.clcc.2014.12.007. Epub 2014 Dec 31. PMID 25677122
- [Background] Ekkarat P, Boonpipattanapong T, Tantiphlachiva K, Sangkhathat S. Factors determining low anterior resection syndrome after rectal cancer resection: A study in Thai patients. Asian J Surg. 2016 Oct;39(4):225-31. doi: 10.1016/j.asjsur.2015.07.003. Epub 2015 Sep 2. PMID 26340884
- [Background] Gadan S, Floodeen H, Lindgren R, Matthiessen P. Does a Defunctioning Stoma Impair Anorectal Function After Low Anterior Resection of the Rectum for Cancer? A 12-Year Follow-up of a Randomized Multicenter Trial. Dis Colon Rectum. 2017 Aug;60(8):800-806. doi: 10.1097/DCR.0000000000000818. PMID 28682965
- [Background] Greimel E, Bottomley A, Cull A, Waldenstrom AC, Arraras J, Chauvenet L, Holzner B, Kuljanic K, Lebrec J, D'haese S; EORTC Quality of Life Group and the Quality of Life Unit. An international field study of the reliability and validity of a disease-specific questionnaire module (the QLQ-OV28) in assessing the quality of life of patients with ovarian cancer. Eur J Cancer. 2003 Jul;39(10):1402-8. doi: 10.1016/s0959-8049(03)00307-1. PMID 12826043
- [Background] Harpain F, Kranawetter M, Zott T, Lazaridis II, Guenin MO, Ninkovic M, Kronberger IE, Tapiolas I, Basany EE, Dauser B, Herbst F, Koh C, Stift A, Teleky B, Reinthaller A, Grimm C, Riss S. Low anterior resection syndrome (LARS) in ovarian cancer patients - A multi-centre comparative cohort study. Int J Surg. 2020 Jun;78:97-102. doi: 10.1016/j.ijsu.2020.04.019. Epub 2020 Apr 15. PMID 32304899
- [Background] Kim CW, Jeong WK, Son GM, Kim IY, Park JW, Jeong SY, Park KJ, Lee SH. Validation of Korean Version of Low Anterior Resection Syndrome Score Questionnaire. Ann Coloproctol. 2020 Apr;36(2):83-87. doi: 10.3393/ac.2019.08.01. Epub 2020 Feb 11. PMID 32054239
- [Background] Kim MJ, Park JW, Lee MA, Lim HK, Kwon YH, Ryoo SB, Park KJ, Jeong SY. Two dominant patterns of low anterior resection syndrome and their effects on patients' quality of life. Sci Rep. 2021 Feb 11;11(1):3538. doi: 10.1038/s41598-021-82149-9. PMID 33574345
- [Background] Kranawetter M, Ataseven B, Grimm C, Schneider S, Riss S, Alesina P, Prader S, Walz MK, Harpain F, Stift A, Heitz F, Reinthaller A, Polterauer S, Harter P, du Bois A. Low anterior resection syndrome (LARS) in patients with epithelial ovarian cancer after primary debulking surgery. Gynecol Oncol. 2019 Sep;154(3):577-582. doi: 10.1016/j.ygyno.2019.06.015. Epub 2019 Jun 21. PMID 31235241
- [Background] Park SJ, Mun J, Lee EJ, Park S, Kim SY, Lim W, Song G, Kim JW, Lee S, Kim HS. Clinical Phenotypes of Tumors Invading the Rectosigmoid Colon Affecting the Extent of Debulking Surgery and Survival in Advanced Ovarian Cancer. Front Oncol. 2021 Apr 22;11:673631. doi: 10.3389/fonc.2021.673631. eCollection 2021. PMID 33968784
- [Background] Rockwood TH, Church JM, Fleshman JW, Kane RL, Mavrantonis C, Thorson AG, Wexner SD, Bliss D, Lowry AC. Patient and surgeon ranking of the severity of symptoms associated with fecal incontinence: the fecal incontinence severity index. Dis Colon Rectum. 1999 Dec;42(12):1525-32. doi: 10.1007/BF02236199. PMID 10613469
- [Background] Rockwood TH, Church JM, Fleshman JW, Kane RL, Mavrantonis C, Thorson AG, Wexner SD, Bliss D, Lowry AC. Fecal Incontinence Quality of Life Scale: quality of life instrument for patients with fecal incontinence. Dis Colon Rectum. 2000 Jan;43(1):9-16; discussion 16-7. doi: 10.1007/BF02237236. PMID 10813117
- [Background] Shimada M, Kigawa J, Minagawa Y, Irie T, Takahashi M, Terakawa N. Significance of cytoreductive surgery including bowel resection for patients with advanced ovarian cancer. Am J Clin Oncol. 1999 Oct;22(5):481-4. doi: 10.1097/00000421-199910000-00012. PMID 10521063
- [Background] Son JH, Kim J, Shim J, Kong TW, Paek J, Chang SJ, Ryu HS. Comparison of posterior rectal dissection techniques during rectosigmoid colon resection as part of cytoreductive surgery in patients with epithelial ovarian cancer: Close rectal dissection versus total mesorectal excision. Gynecol Oncol. 2019 May;153(2):362-367. doi: 10.1016/j.ygyno.2019.02.029. Epub 2019 Mar 4. PMID 30846223
- [Background] Yun YH, Park YS, Lee ES, Bang SM, Heo DS, Park SY, You CH, West K. Validation of the Korean version of the EORTC QLQ-C30. Qual Life Res. 2004 May;13(4):863-8. doi: 10.1023/B:QURE.0000021692.81214.70. PMID 15129896